CLINICAL TRIAL: NCT01739803
Title: Behavioral Contract Intervention to Improve Adherence Among Renal Transplant Recipients
Brief Title: Behavioral Contract Adherence Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7R01DK081347-04 (NIH); 7R01DK081347-04 (NIH)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2013-12

CONDITIONS: Renal Transplantation
Keywords: Immunosuppressant therapy adherence; Quality of life; Economic outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Behavioral contract intervention
  Interventions: Behavioral: Behavioral Contract
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Behavioral Contract — Intervention activities were performed by a study clinical pharmacist. Behavioral contract goal was achieving and maintaining IST adherence. Other components of the contract addressed: (a) motivation(s) or positive reinforcement for achieving IST adherence; (b) problems or barriers that may interfere with achieving IST adherence and possible solutions to overcome problems/barriers; (c) social support available to the RTR such as a significant other who may assist the RTR in following the IST dosing schedule; (d) tools/strategies the RTR may use to remind himself/herself to follow the IST dosing schedule; and (e) possible consequences of IST nonadherence (e.g., graft loss).
  Arms: Intervention Group

SUMMARY:
There is a critical gap in the knowledge on how to implement effective interventions for renal transplant recipients (RTRs) to improve immunosuppressant therapy (IST) adherence and clinical outcomes. The objectives of this project were to address this gap through: (1) designing, implementing, and evaluating a patient-specific behavioral contract intervention to improve RTRs' IST adherence rates (contracts are written, signed agreements between the RTR and healthcare provider in which the RTR agrees to be adherent to IST according to mutually agreed upon criteria); and (2) measuring the effects of IST adherence on RTRs' health-related quality of life (HQoL) and healthcare utilizations and costs. The primary hypothesis was that at one year post trial enrollment, RTRs who establish behavioral contracts with healthcare professionals will be more adherent than those who do not establish behavioral contracts and subsequently will have greater HQoL and lower healthcare utilizations and costs. Once it is better understood how to implement effective IST adherence intervention programs, clinicians will have a valuable tool to promote therapeutic success, improve HQoL, and reduce healthcare utilizations and costs. Therefore, we pursued the following Specific Aims: (1) determine the effectiveness of an IST adherence contract-based intervention on IST adherence; (2) determine the relationship between IST adherence, the intervention, and RTRs' HQoL; and (3) determine the influence of IST adherence and the intervention on RTRs' healthcare utilizations/costs. To achieve the Specific Aims, a randomized controlled trial of the patient-specific behavioral contract-based intervention was conducted, and data regarding adherence, HQoL, and healthcare utilizations/costs were collected over a 12-month period for each RTR study participant and analyzed. This project will promote healthy lives, increase well-being, and reduce burden of illness and disparity among adult RTRs by providing data regarding an adherence intervention and the impact of IST adherence and the behavioral contract intervention on RTRs' health and economic outcomes and HQoL. Collectively, this new knowledge will provide critical steps toward optimizing RTRs' graft maintenance, productivity, and HQoL, while decreasing graft rejection, return to dialysis, morbidity, mortality, and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipient
* at least 21 years of age
* receive an immunosuppressant regimen that contains oral cyclosporine or tacrolimus
* be at least one year post-transplant
* obtain immunosuppressant therapy from Avella Specialty Pharmacy for at least one year prior to study enrollment and during the study period

Exclusion Criteria:

* pregnant
* prisoner
* institutionalized
* unable to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Chisholm-Burns, PharmD, Principal Investigator — University of Tennessee College of Pharmacy
Locations (1):
- University of Arizona College of Pharmacy, Tucson, Arizona, United States

REFERENCES:
- [Background] Chisholm-Burns MA, Erickson SR, Spivey CA, Gruessner RW, Kaplan B. Concurrent validity of kidney transplant questionnaire in US renal transplant recipients. Patient Prefer Adherence. 2011;5:517-22. doi: 10.2147/PPA.S24261. Epub 2011 Oct 13. PMID 22114465
- [Background] Chisholm-Burns MA, Erickson SR, Spivey CA, Kaplan B. Health-related quality of life and employment among renal transplant recipients. Clin Transplant. 2012 May-Jun;26(3):411-7. doi: 10.1111/j.1399-0012.2011.01541.x. Epub 2011 Oct 28. PMID 22032257
- [Result] Chisholm-Burns MA, Spivey CA, Graff Zivin J, Lee JK, Sredzinski E, Tolley EA. Improving outcomes of renal transplant recipients with behavioral adherence contracts: a randomized controlled trial. Am J Transplant. 2013 Sep;13(9):2364-73. doi: 10.1111/ajt.12341. Epub 2013 Jul 2. PMID 23819827
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: RTRs were enrolled between January 2010 and September 2011 and followed for one year (the study or intervention period). All active participants completed the study by September 2012; however, refill records were collected for three months following the end of the study period to calculate a follow-up (post-intervention) adherence rate.
Pre-assignment Details: Inclusion criteria: (a) at least 21 years of age; (b) at least one year post-transplant to allow for stabilization of the prescribed IST regimen; (c) receive an immunosuppressant regimen that contains oral tacrolimus or cyclosporine; and (d) obtain their IST from Avella for at least one year prior to study enrollment and during the study period.
Groups:
- Intervention Group: Behavioral contract intervention.
  Each participant in the intervention group met with the study pharmacist to negotiate and sign an immunosuppressant therapy (IST) adherence contract at baseline. Each intervention participant met with the study pharmacist at 3-, 6-, and 9-months post-enrollment to review his or her contract, discuss progress toward reaching the contract's goal of achieving the highest possible IST adherence, update terms of the contract if needed, and re-sign the contract for the next three-month period. At the 12-month post-enrollment meeting, the contract was terminated.
  The contract included: (a) motivation(s) for achieving adherence; (b) barriers that may interfere with achieving adherence and possible solutions to overcome barriers; (c) social support available such as a significant other who may assist in following the dosing schedule; (d) tools/strategies to follow the dosing schedule; and (e) possible consequences of nonadherence
- Control Group: No intervention.
  The control group received standard specialty pharmacy care, which included mail or telephone reminders of monthly medication refills and an adherence "packet" consisting of adherence-focused educational pamphlets and a pillbox
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 76 | 74
Completed | 67 | 68
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 62 | 121
  >=65 years | 17 | 12 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.78 (13.55) | 51.32 (13.69) | 52.06 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 43 | 41 | 84
Region of Enrollment [Number; unit: participants]
  United States | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Average Immunosuppressant Therapy Adherence for 12-month Study Period
Description: Immunosuppressant therapy adherence as measured by pharmacy refill records. Adherence was calculated quarterly for one year by using the number of days between prescription (IST) refills. If the total number of days between refills was less than or equal to the total days' supply of IST, the participant's adherence rate was 1.0, or 100%. If the number of days between refills was greater than the days' supply, the adherence rate was calculated as follows:
  1 - [(Days Between Refills - Total Days Supply)/Days Between Refills] = Adherence Rate for Quarterly Time Period
  At the end of the 12-month study period, the quarterly adherence rates were averaged to produce an overall adherence rate for the study period.
Time Frame: 12 months
Population: Intention to treat, as per protocol
Measure: Mean (Standard Deviation); unit: medication possession ratio (proportion)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 76 | 74
medication possession ratio (proportion) | 0.88 (0.17) | 0.81 (0.18)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We projected mean composite adherence rate for all participants to be approximately 80% ± 15. We anticipated at least 10% increase in intervention group adherence at end of intervention. To have 80% power to detect expected difference of 10% at the 2-tailed 5% significance level, sample size needed to be at least 36 RTRs per group. We took a conservative approach, in combination with anticipated attrition over the course of study, and increased enrollment; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — To control for experiment-wise Type I error rate in this analysis, a comparison-wise alpha of 0.01 was used

2. Secondary Outcome: Health-related Quality of Life (HQoL)
Description: The EQ-5D is a multi-attribute, preference-based HQoL instrument. Considered a global HQoL measure, the EQ-5D is a descriptive system that classifies respondents into one of 243 distinct health states based on five dimensions (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has three levels, reflecting "no problems," "some problems," and "extreme problems." A scoring function assigns a value (EQ-5DIndex score) to self-reported health states from a set of preference weights that have been empirically derived. The EQ-5D's total scale (preference value) range is from 0 to 1.0. On this scale, the preference value of 1.0 represents perfect health and 0.0 represents death. Preference values less than 0 are possible, but not reflected on the scale, and reflect health states that the U.S. population consider worse than death.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 68
units on a scale | 0.84 (0.17) | 0.85 (0.18)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.05, ANOVA

3. Secondary Outcome: Days in Hospital
Description: We used a standardized patient reporting approach to collect direct healthcare utilizations data, including days in hospital. A brief healthcare screening questionnaire was administered to both the intervention and control groups on a monthly basis during the one-year study period. Monthly recall periods were chosen to minimize bias and forgetfulness. The questionnaire collected the number of times each month a participant utilized a direct medical service, specifically, days in hospital, emergency department (ED) visit, outpatient visit (clinic, physician office), and home healthcare visit.
  Analysis compared proportion of each group who had at least one day in hospital during the 12-month study period.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 67 | 68
percentage of participants | 51 (0.22) | 29 (0.99)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.05

ADVERSE EVENTS:
Time Frame: 12 month study period
Description: No risks were anticipated as intervention participants received support (behavioral contract) to take medication as prescribed and control group received standard care.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/74

LIMITATIONS AND CAVEATS:
Did not include attention control group. Did not employ multiple study pharmacists to perform intervention. Limitations of pharmacy refill records: accuracy may be affected by dosage changes, do not indicate if drug actually consumed as prescribed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No